CLINICAL TRIAL: NCT00901225
Title: Plerixafor Rescue Mobilization For Autologous Stem Cell Transplant Patients With Inadequate Response to G-CSF
Brief Title: Study of Plerixafor for Rescue of Poor Mobilizers in Autologous Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014563
Record Dates: First submitted 2009-05-04; First posted 2009-05-13 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Myeloma; Non-Hodgkins Lymphoma; Hodgkins Disease
Keywords: NHL
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- G-CSF plus Plerixafor (Experimental): Patients who were unable to mobilize a minimum number of cells (CD34+ cell count <20 cells/ul)following 5 days of G-CSF mobilization.
  Interventions: Drug: G-CSF plus Plerixafor

INTERVENTIONS:
Drug: G-CSF plus Plerixafor — On Day 5 of G-CSF mobilization,
  1. if the patient's peripheral CD34+ cell count is < 7cells/µl then 240ug/kg Plerixafor will be given in the evening prior to receiving 10µg/kg G-CSF and undergoing apheresis the next morning for up to 3 days of apheresis or until ≥ 5x10(6) cells/kg are collected.
  2. if the patient's peripheral CD34+ cell count is 7 to 19 cells/ul (inclusive), apheresis will be done. If the apheresis yield is < 1.3x10(6) CD34+ cells/kg then 240ug/kg Plerixafor will be given in the evening prior to receiving 10 µg/kg G-CSF and undergoing apheresis the next morning. If the apheresis yield is at least double that on Day 5, Plerixafor followed the next morning by G-CSF and apheresis will be repeated for up to a total of 3 days of apheresis or until 5x10(6) cells/kg are collected.
  Other Names: Mozobil, AMD3100

SUMMARY:
Plerixafor, administered at a dose of 240 ug/kg, potentiates the effect of granulocyte colony-stimulating factor (G-CSF) to increase peripheral blood progenitor cells in both healthy volunteers and cancer patients. Furthermore, in cancer patients, cells collected via apheresis using Plerixafor and G-CSF have been successfully transplanted. In December 2008, Plerixafor received approval from the Food and Drug administration for use in combination with G-CSF to aid in mobilization of progenitor cells for apheresis. The proposed study is not designed to support approval of a new indication or change in the advertising for Plerixafor. The route of administration and dosage level are identical to that which is listed on the package insert. Although Plerixafor is not approved for patients with Hodgkins Lymphoma, there is no known or theoretic increased risk of the use of this drug in this patient population.

The study hypothesis for this study is that patients with a circulating CD34+ count < 20 cells/ul after 5 days of mobilization with G-CSF alone will achieve > or equal to 2 X 10(6)CD34+ cells/kg within 3 days of apheresis after receiving Plerixafor with G-CSF.

DETAILED DESCRIPTION:
This is a single-center, Phase 2, open-label study. All patients diagnosed with non-hodgkins lymphoma, hodgkins disease or multiple myeloma and candidates for autologous transplantation are eligible to enter into the study. The only change to the standard of care is the addition of 240 ug/kg Plerixafor following 5 days of (G-CSF) mobilization.

The results of the study will provide both numeric and categorical estimates of measurements of the safety and efficacy of Plerixafor. The primary efficacy endpoint, Treatment Success, is a binary response variable categorizing whether the patient was able to mobilize at least 2 X 10(6) CD34+ cells/kg within 3 days of apheresis.

The percentage of patients achieving Treatment Success will be summarized. All AEs will be followed for 30 days after the last apheresis or until the first dose of ablative chemotherapy, whichever occurs first. All SAEs will be followed for 6 months post-transplant or until relapse. All patients who receive at least one dose of Plerixafor will be included in all summaries of AEs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years.
* Diagnosis of NHL, HD or MM
* Eligible for autologous transplantation
* CD34+ cell count < 7 cells/ul after 5 days of mobilization with G-CSF or CD34+ cell count between 7 and 19 (inclusive) on day 5 of mobilization with G-CSF and < 1.3 x 106 CD34+ cells collected by apheresis on day 5 of G-CSF therapy.
* < or equal to 5 prior regimens of chemotherapy (Rituxan is not considered chemotherapy for the purpose of this study)
* ≥ 3 weeks since last cycle of chemotherapy and the beginning of G-CSF mobilization (Rituxan and Lenalidomide are not considered chemotherapy for the purpose of this study)
* Total dose of melphalan < or equal to 200 mg
* ECOG performance status of 0 or 1
* Recovered from all acute toxic effects of prior chemotherapy
* Absolute PMN count > 1.0 X 10(9)/l prior to first dose of G-CSF
* PLT count > 75 X 10(9)/l prior to first dose of G-CSF
* Serum creatinine < or equal to 2.5 mg/dl
* SGOT, SGPT and total bilirubin < 2 X upper limit of normal (ULN) prior to the first dose of G-CSF
* Cardiac and pulmonary status sufficient to undergo apheresis and transplantation as determined by standard institutional practice
* Signed informed consent
* Patients of childbearing potential agree to use an approved form of contraception

Exclusion Criteria:

* A co-morbid condition which, in the view of the investigator, renders the patient at high risk from treatment complications
* Failed previous stem cell collection or collection attempts
* A residual acute medical condition resulting from prior chemotherapy
* Active brain metastases or carcinomatous meningitis
* Active infection requiring antibiotic treatment (excluding controlled catheter-related bacteremia)
* Received prior radio-immunotherapy with Zevalin or Bexxar
* Received thalidomide, dexamethasone, and/or Velcade within 7 days prior to the first dose of G-CSF
* Positive pregnancy test in female patients
* Lactating females
* Patients who previously received experimental therapy within 4 weeks of enrolling in this protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled in April 2005 and the final patient enrolled in August 2010. The protocol was closed to accrual for approximately 3.5yrs, so the total time to protocol activation was 15 months. This was a single institution study (Duke adult stem cell transplant program).
Pre-assignment Details: All patients deemed to be poor mobilizers to G-CSF as a single agent, were eligible for enrollment (assuming protocol eligibility criteria were met).
Period: Overall Study
Arm/Group | G-CSF Plus Plerixafor
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | G-CSF Plus Plerixafor
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved > or Equal to 2 X 10(6)CD34+ Cells/kg Within 3 Days of Apheresis After Receiving Plerixafor With G-CSF.
Time Frame: 5 days after receiving G-CSF
Measure: Number; unit: participants
Arm/Group | G-CSF Plus Plerixafor
Number analyzed (Participants) | 20
participants | 15

2. Secondary Outcome: Number of Participants Experiencing a Grade III/IV Toxicity
Description: Safety of plerixafor as measured by Grade III/IV Toxicity
Time Frame: 6 months post transplant or until relapse
Measure: Number; unit: participants
Arm/Group | G-CSF Plus Plerixafor
Number analyzed (Participants) | 20
participants | 0

3. Secondary Outcome: Number of Subjects Experiencing Graft Failure
Description: To investigate the hematological activity of Plerixafor as measured by Graft Failure. Graft failure is defined as failure of initial engraftment (primary graft failure) or initial engraftment, but subsequent loss of hematopoiesis (secondary graft failure).
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | G-CSF Plus Plerixafor
Number analyzed (Participants) | 20
participants | 0

4. Secondary Outcome: Days to Absolute Neutrophil Count >500
Time Frame: 12 months
Measure: Median (Full Range); unit: days
Arm/Group | G-CSF Plus Plerixafor
Number analyzed (Participants) | 20
days | 11 [10 to 16]

5. Secondary Outcome: Number of Subjects Experiencing Durability of Engraftment
Description: Durability of engraftment is defined as the duration and stability of hematopoiesis following autologous transplantation. Subjects who experience durable engraftment have neutrophil counts greater than 500 and platelet counts greater than 20,000 within the specified time frame.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | G-CSF Plus Plerixafor
Number analyzed (Participants) | 20
participants | 20

6. Secondary Outcome: Platelet Engraftment
Description: Days to platelet count >20,000
Time Frame: 12 months
Measure: Median (Full Range); unit: days
Arm/Group | G-CSF Plus Plerixafor
Number analyzed (Participants) | 20
days | 19 [10 to 44]

ADVERSE EVENTS:
Arm/Group | G-CSF Plus Plerixafor
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 4/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-CSF Plus Plerixafor (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (6) — fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No